CLINICAL TRIAL: NCT05493995
Title: A Multicenter Study of Penpulimab and Anlotinib in Combination With Nab-paclitaxel Plus Gemcitabine as First-line Therapy in Patients (Pts) With Metastatic Pancreatic Cancer: PAAG.
Brief Title: A Study of Penpulimab and Anlotinib Plus Nab-paclitaxel and Gemcitabine for Metastatic Pancreatic Cancer.
Acronym: PAAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Du Juan, Clinical Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-351-02
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — penpulimab; anlotinib; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab+Anlotinib+Nab-paclitaxel+Gemcitabine (Experimental)
  Interventions: Drug: Penpulimab; Drug: Anlotinib; Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Penpulimab — Penpulimab 200 mg administered intravenously every 3 weeks.
  Other Names: AK105
Drug: Anlotinib — 12mg, continuous oral 2 weeks stop for 1 week, 21 days for a treatment cycle.
Drug: Nab paclitaxel — 125mg/m^2，administered intravenously on days 1 and 8 of every 21-day cycle.
Drug: Gemcitabine — 1.0g/m^2, administered intravenously on days 1 and 8 of every 21-day cycle.

SUMMARY:
It is a trial to assess the efficacy and safety of Penpulimab and Anlotinib in Combination With Nab-paclitaxel Plus Gemcitabine as first-line Therapy in Patients (Pts) With Metastatic Pancreatic Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥18 years，ECOG ≤ 2，Estimated survival time > 3 months
* Histologically or Cytologically confirmed metastatic pancreatic adenocarcinoma
* Based on Response Evaluation Criteria In Solid Tumors (RECIST1.1), there should be at least one measurable lesion
* Patients have never received systematical anti-cancer therapy
* Laboratory examination meets the following requirements:White blood cell (WBC) ≥3.0×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; Hemoglobin (HB) ≥90g/L; platelet count(PLT) ≥75×109/L; Total bilirubin (TBIL) ≤1.5× normal upper limit (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST)≤2.5×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN; Serum creatinine (Cr) ≤1×ULN or creatinine clearance (CCr)≥50ml/min;
* Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) > 50%
* Patients of childbearing age should take appropriate protective measures before enrollment and during the trial
* Volunteer to join the study, sign the informed consent, have good compliance, and cooperate with follow-up
* Ability to follow the study protocol and follow-up procedures.

Exclusion Criteria:

* Patients have ever received any systematical anti-cancer therapy in the past
* Patients who participated in other clinical trials in the past 4 weeks
* According to the investigator, patients who surgically available or potentially treatable(Patients who voluntarily give up surgical treatment can be enrolled after evaluation by the investigator)
* Patients with moderate ascites requiring drainage
* Patients with CNS metastases and/or carcinomatous meningitis
* Patients with history of other primary malignancies except: 1) complete remission before enrollment for at least 2 years and requiring no additional treatment during the study period; 2) Adequately treated non-melanoma skin cancer or lentiform malignancy with no evidence of disease recurrence; 3) Adequately treated carcinoma in situ with no evidence of disease recurrence;
* Patients with autoimmune disease or immune deficiency who are treated with immunosuppressive drugs
* Patients with bleeding tendency.
* Pregnant or lactating women.
* Drug abuse, clinical or psychological or social factors that impact informed consent or the conduct of the study
* Patients who may be allergic to PD-1 monoclonal antibody, anlotinib, albumin-bound paclitaxel and gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 3 years
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the Response Evaluation Criteria In Solid Tumors Criteria(RECIST v1.1).
Disease Control Rate (DCR) | up to 3 years
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 3 years
  Overall Survival (OS) (median) is determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.
Progression-free survival (PFS) | up to 3 years
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Sha H, Tong F, Ni J, Sun Y, Zhu Y, Qi L, Li X, Li W, Yang Y, Gu Q, Zhang X, Wang X, Zhu C, Chen D, Liu B, Du J. First-line penpulimab (an anti-PD1 antibody) and anlotinib (an angiogenesis inhibitor) with nab-paclitaxel/gemcitabine (PAAG) in metastatic pancreatic cancer: a prospective, multicentre, biomolecular exploratory, phase II trial. Signal Transduct Target Ther. 2024 Jun 7;9(1):143. doi: 10.1038/s41392-024-01857-6. PMID 38844468